CLINICAL TRIAL: NCT06157788
Title: Cerebral Activation Related to Shoulder Apprehension in Patients With Glenohumeral Instability. A Concise Follow-up of a Previous Report.
Brief Title: Cerebral Activation and Apprehension in Patients With Shoulder Instability.
Status: Completed | Type: Observational
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Dr. Alexandre Lädermann, Orthopaedic Surgeon, La Tour Hospital
Other Study IDs: 2022-00135
Record Dates: First submitted 2023-11-27; First posted 2023-12-06 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Shoulder Instability
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operated group: Patients were male individuals with anterior glenohumeral instability, who underwent preoperative fMRI, then surgical stabilization by 2 specialized shoulder surgeons, followed by a new fMRI one year postoperatively.
  Interventions: Diagnostic Test: functional Magnetic Resonance Imaging and clinical assessment
- Control Group: The control group consisted in healthy volunteers with no history of shoulder injury, instability, or hyperlaxity, the latter defined as more than 85° of external rotation elbow against waist, or hyperabduction over 105°, who had undergone fMRI at baseline.
  Interventions: Diagnostic Test: functional Magnetic Resonance Imaging and clinical assessment

INTERVENTIONS:
Diagnostic Test: functional Magnetic Resonance Imaging and clinical assessment — * fMRI task: In the active condition, video cues were utilized (lasting 10s) depicting everyday activities that trigger shoulder apprehension. Control videos were created to match the previous content, except for the absence of cues inducing shoulder apprehension. Following each video, a visual analog scale appeared for a duration of 2.5s, and participant were asked to rate the level of perceived apprehension, using an MRI-compatible response box. The rating scale consisted of nine steps, ranging from no apprehension to high apprehension. After providing their rating, participants had a rest period during which a fixation cross was displayed visually for 17.5s. Apprehension and control videos were shown in a pseudo-randomized fashion.
  * General Linear Model Analysis of Task-Related Activation
  * TICA Analysis of Functional Connectivity
  * White Matter TBSS of DTI Data
  * Voxel-based morphometry analysis of T1 images

SUMMARY:
In a similar study, the investigators demonstrated that shoulder stabilization could allow the brain to partially "recover". Patients with shoulder apprehension underwent clinical and fMRI examination before and one year after shoulder stabilization surgery. Clinical examination showed a significant improvement in postoperative shoulder function compared with preoperative. Coherently, results showed a decreased activation in the left pre-motor cortex postoperatively, demonstrating that stabilization surgery induced improvements both at the physical and at the brain levels, one year postoperatively. Most interestingly, right-frontal pole and right-occipital cortex activity was associated with good outcome in shoulder performance.

DETAILED DESCRIPTION:
Fear, anxiety and anticipation of situations that could lead to a dislocation are essential cognitive processes in shoulder apprehension. Functional magnetic resonance imaging (fMRI) measures brain activity by detecting changes associated with blood flow. This technique relies on the fact that cerebral blood flow and neuronal activation are coupled. When an area of the brain is in use, blood flow to that region also increases. Recently, investigators used fMRI with visual apprehension stimulation to explore neuronal connections and cerebral changes induced by shoulder dislocation. Several cerebral areas were modified during those analyses, representing the different aspects of shoulder apprehension. Specific reorganizations were found in apprehension-related functional connectivity of the primary sensory-motor areas (motor resistance), dorsolateral prefrontal cortex (cognitive control of motor behavior), and the dorsal anterior cingulate cortex/dorsomedial prefrontal cortex and anterior insula (anxiety and emotional regulation).

Those regions are involved in the cognitive control of motor behavior. Hence, there is a motor control anticipation and muscular resistance (protective reflex mechanism), in order to avoid shoulder movement that could lead to dislocation. Another recent study published by Shitara et al. analyzed cerebral changes induced by shoulder dislocation in 14 patients. Although results were similar to the investigators' study, they observed a larger and less specific spectrum of activated cerebral areas, that may be explained by the fact that they projected static and abstract images during fMRI acquisition that may be prone to vaguer and subjective interpretation, and that moreover did not convey the dynamic component inherent to apprehension. In a subsequent study, investigators extended these findings by investigating further structural alterations in patients with shoulder apprehension. The investigators found that fractional anisotropy, representing white matter integrity, was increased in the left internal capsule and partially in the thalamus of studied patients compared to healthy controls. Fractional anisotropy correlated positively with pain visual analogue scale (VAS) scores (p < .05) and negatively with simple shoulder test (SST) scores (p < .05). This suggests an abnormal increased axonal integrity and therefore pathological structural plasticity due to the over-connection of white matter fibers in the motor pathway. These structural alterations affect several dimensions of shoulder apprehension as pain perception and performance in daily life.

The neuronal changes previously mentioned and presented in shoulder apprehension can also be assessed in daily clinical practice. Indeed, Cunningham et al. correlated clinical scores and tests (Rowe, pain VAS, SST, subjective shoulder value (SSV), WOSI) with functional cerebral imaging in patients with shoulder apprehension. Their hypothesis was that it might be possible to simplify shoulder instability scores as it has been previously possible with rotator cuff and SLAP lesions, and that at least one score could encompass the spectrum of these cerebral alterations. They found that the Rowe score integrated several aspects of apprehension, notably the motor and sensory functions, as well as pain anticipation and attention. This could be explained by the fact that the Rowe score is the only tested score that integrates range of motion. This also provides the ability to evaluate motor component (stability and motion) and cognitive component (perceived pain) of shoulder apprehension. Pain VAS and WOSI seemed to correlate with less brain networks compared to the Rowe. This could be explained by the fact that their assessment is focused only on cognitive aspects (pain for pain VAS, shoulder function in everyday life activities for WOSI), and that they do not integrate pure shoulder motion. SST and SSV were not found to be associated with brain network alterations, which is corroborated by the fact that they are general shoulder scores and were not specifically validated for instability.

In a similar study, the investigators demonstrated that shoulder stabilization could allow the brain to partially "recover". Patients with shoulder apprehension underwent clinical and fMRI examination before and one year after shoulder stabilization surgery. Clinical examination showed a significant improvement in postoperative shoulder function compared with preoperative. Coherently, results showed a decreased activation in the left pre-motor cortex postoperatively, demonstrating that stabilization surgery induced improvements both at the physical and at the brain levels, one year postoperatively. Most interestingly, right-frontal pole and right-occipital cortex activity was associated with good outcome in shoulder performance.

ELIGIBILITY:
Inclusion Criteria:

* The 15 patients operated 10 years ago and the 15 patients used as a control group in a previous analysis.

Exclusion Criteria:

* Previous recurrence of instability reported in the past 10 years.
* Major medical disorders (cancer, cardiac illness)
* Sustained head injury
* Psychiatric or neurologic disorders
* Alcohol or drug abuse
* Use of psychotropics, stimulants, and beta-blockers on a regular basis
* Abnormal or non-corrected-to-normal visual acuity
* New contra-indication for fMRI, such as claustrophobia, pacemaker

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients were male individuals with anterior glenohumeral instability, who underwent preoperative fMRI, then surgical stabilization by 2 specialized shoulder surgeons, followed by a new fMRI one year postoperatively. The control group consisted in healthy volunteers with no history of shoulder injury, instability, or hyperlaxity, the latter defined as more than 85° of external rotation elbow against waist, or hyperabduction over 105°, who had undergone fMRI at baseline.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Task-related brain activation | At 10 post-operative years
  Temporal independent component analysis of functional Connectivity

SECONDARY OUTCOMES:
Behavioural responses to apprehension videos | At 10 post-operative years
  Minimum 1 (No Apprehension), Maximum 7 (Apprehension)
Changes in grey matter | At 10 post-operative years
  Structural changes in grey matter using voxel-based morphometry
Changes in white matter | At 10 post-operative years
  structural changes in white matter using tract-based spatial statistics analysis with multimodal Magnetic Resonance imaging
Pain on visual analog scale | At 10 post-operative years
  From 0 (no pain) to 10 (extreme pain)
Subjective Shoulder Value | At 10 post-operative years
  SSV (Subjective Shoulder Value). From 0 (worst) to 100 (best)
Rowe score | At 10 post-operative years
  From 0 (worst) to 100 (best)
Simple Shoulder Test | At 10 post-operative years
  From 0 (worst) to 12 (best)
Western Ontario Shoulder Instability Index | At 10 post-operative years
  From 0 (worst) to 100 (best)
Single Assessment numeric evaluation score | At 10 post-operative years
  Single Assessment numeric evaluation (SANE). From 0 (worst) to 100 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- La Tour hospital, Meyrin, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Haller S, Cunningham G, Laedermann A, Hofmeister J, Van De Ville D, Lovblad KO, Hoffmeyer P. Shoulder apprehension impacts large-scale functional brain networks. AJNR Am J Neuroradiol. 2014 Apr;35(4):691-7. doi: 10.3174/ajnr.A3738. Epub 2013 Oct 3. PMID 24091445